CLINICAL TRIAL: NCT00562549
Title: A Pilot Phase IIa Randomised, Double-blind, Placebo-controlled, Crossover Study to Examine the Safety, Tolerability and Pharmacodynamic Effects on Blood Pressure of Repeat Oral Doses of SLx-2101 5, 10 or 20 mg Once Daily for up to 14 Days in Patients With Hypertension
Brief Title: Safety and Effects of SLx-2101 Taken for up to 14 Days on Blood Pressure in Patients With Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Response Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SLx-2101-07-05
Record Dates: First submitted 2007-11-20; First posted 2007-11-22 (Estimated); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): SLx-2101
  Interventions: Drug: SLx-2101
- 2 (Placebo Comparator): Matching Placebo Dose
  Interventions: Drug: SLx-2101

INTERVENTIONS:
Drug: SLx-2101

SUMMARY:
The purpose is to determine the effective dosage and to study the effects of this dosage taken for 12 days on systolic and diastolic blood pressure in patients with hypertension.

DETAILED DESCRIPTION:
1. Office seated peripheral systolic and diastolic blood pressure
2. Adverse events and vital signs
3. Plasma concentrations of SLx-2101

ELIGIBILITY:
Inclusion Criteria:

* Male or females between 18 and 80 years, inclusive
* Moderate to severe hypertension
* Body weight within a body mass index range of 18 - 32 kg/m2

Exclusion Criteria:

* Subject is receiving more than four antihypertensive agents
* History of drug abuse
* Exposure to a new chemical entity within 3 months prior to the first day of dosing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Office seated peripheral systolic and diastolic blood pressure | 12 days

SECONDARY OUTCOMES:
Adverse events and changes in vital signs | 12 days

CONTACTS AND LOCATIONS:
Overall Officials: Ian B Wilkinson, MD, Principal Investigator — Addenbrooke's Hospital, Cambridge
Locations (1):
- Addenbrooke's Hospital, Cambridge, United Kingdom